CLINICAL TRIAL: NCT04747717
Title: Efficacy of Neoadjuvant Therapy With Cisplatin Plus Mitomycin C in BRCA1-Mutated Ovarian Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: N.N. Petrov National Medical Research Center of Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OvCa-NeoMP
Record Dates: First submitted 2021-01-29; First posted 2021-02-10 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-01

CONDITIONS: Ovarian Cancer
Keywords: Ovarian cancer; Neoadjuvant chemotherapy; Mitomycin C
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Drug Therapy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mitomycin C and cisplatin regimen (Experimental): mitomycin C at 10 mg/m2 and cisplatin at 100 mg/m2
  Interventions: Procedure: chemotherapy/surgery
- Paclitaxel and carboplatin regimen (Active Comparator): paclitaxel at 175 mg/m2 and carboplatin AUC5-6
  Interventions: Procedure: chemotherapy/surgery

INTERVENTIONS:
Procedure: chemotherapy/surgery — NEO chemotherapy/interval debulking surgery/AD chemotherapy

SUMMARY:
This study was designed to assess the safety and efficacy of neoadjuvant therapy with mitomycin C plus cisplatin (MP) in BRCA1-mutated ovarian cancer versus standard regimen (paclitaxel plus carboplatin (TP)).

DETAILED DESCRIPTION:
The trial includes two arms, one of which is experimental arm with MP regimen chemotherapy that is compared with other arm with the standard TC regimen chemotherapy. To participate in this study, patients must have histologically confirmed epithelial ovarian carcinoma (ОС) or fallopian tubes carcinoma and FIGO stage IIB, IIC, III, or IV disease and BRCA1/BRCA2 germline mutation. All OC patients before the treatment start are subjected to the testing for BRCA1/BRCA2 mutations cases that are examined by the next-generation sequencing. All BRCA1/2 mutation carriers, who could not be treated by primary debulking surgery owing to extensive tumor spread, are given neoadjuvant chemotherapy. OC patients are randomly assigned to receive the TP regimen (paclitaxel at175 mg/m2 and carboplatin AUC5-6) or the MP regimen (mitomycin C at 10 mg/m2 and cisplatin at 100 mg/m2).

After 3-4 cycles of neoadjuvant chemotherapy, a formal assessment is made and patients are categorized according to the RECIST 1.1 standard. The patients who show partial clinical response or complete clinical response has to be undergoing interval debulking surgery. The patients who show stabilization of the process should continue chemotherapy for up to 6 cycles, followed by an assessment of the treatment (it is possible to continue up to 12 cycles) and a decision on whether to perform interval debulking surgery. Patients categorized as progressed clinically has to finish the protocol treatment and are allowed to receive any secondary treatment at the investigators' discretion. For those patients undergoing interval debulking surgery has to receive further regimens (up to 6 cycles of protocol treatment) without changing chemotherapy regimen. After six cycles of protocol treatment, the patients had to be categorized with regard to their final response status with the use of clinical/radiologic assessment. Patients not showing disease progression at this point could cease all cytotoxic therapy or can receive three additional cycles of protocol treatment.

While on protocol therapy, patients underwent the following procedures: symptom recording and physical examination every 3 weeks, complete blood cell counts weekly for the first two cycles and every 3 weeks thereafter, and laboratory tests of blood and CA 125 measurements on day 1 of each cycle.

Radiologic investigations to document the status of all measurable lesions noted at baseline had to be repeated after three, six, and nine cycles of chemotherapy. Once patients were off the protocol therapy, they were monitored for assessment of disease status every 3 months for 2 years and every 6 months thereafter. Monitoring comprised clinical examination and CA 125 estimation; routine computed tomography scans were not required but were requested if the CA 125 level rose and/or symptoms developed.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed epithelial ovarian carcinoma or fallopian tubes carcinoma
* FIGO stage IIB, IIC, III, or IV disease
* BRCA1/BRCA2 germline mutation

Exclusion Criteria:

* WHO performance status >3
* FIGO early stage
* wt BRCA status
* cytological verification

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Response rate | 4 months after FPFV
  To assess the objective response rate (OR) by RECIST v1.1 2. Pathologic response
Pathomorphological response | 4 months after FPFV
  Pathomorphological response will assess after surgery by Bohm scale
Progression Free Survival | 3 years
  As per RECIST v1.1. progression-free survival (PFS) is the time from date of randomization/start of treatment to the date of event defined as the first documented progression or death due to any cause

SECONDARY OUTCOMES:
Adverse events incidence | Until 30 days after last patient treatment visit
  is defined as the interval between the date last chemotherapy cycle and the date of progression of the disease or death or start of a new therapy without evidence of progression, whichever occurred first

CONTACTS AND LOCATIONS:
Overall Officials: Igor Berlev, Study Chair — National Medical Research Centre of Oncology named after N.N. Petrov
Locations (1):
- NMRC of Oncology named after N.N.Petrov of MoH of Russia, Saint Petersburg, Pesochny-2, St.-Petersburg, Russia